CLINICAL TRIAL: NCT02331433
Title: A Phase 1 Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of APN1125 in Healthy Normal Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of Single Doses of APN1125 in Healthy Normal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CoMentis (Industry)
Collaborators: Alpharmagen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APN1125-001
Record Dates: First submitted 2014-12-26; First posted 2015-01-06 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: 1 (Experimental)
  Interventions: Drug: APN1125
- Placebo Comparator: 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APN1125 — APN1125 orally at ascending doses
  Arms: Experimental: 1
Drug: Placebo — Matching Placebo
  Arms: Placebo Comparator: 2

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of APN1125 when administered as single doses to healthy adult subjects.

DETAILED DESCRIPTION:
The study will consist of 2 parts: (1) a single dose in healthy adult volunteers, (2) effect of food upon pharmacokinetics of a single dose of APN1125 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Aged 18 to 65 years, inclusive
* Body mass index (BMI) of 18 to 32kg/m^2 inclusive at Screening
* Non-smoker or no tobacco/nicotine usage with 30 days of Screening

Exclusion Criteria:

* Personal or family history of neurological, cardiovascular, renal, hepatic, metabolic, gastrointestinal or endocrine abnormalities
* Any clinical abnormality in cardiovascular (e.g., blood pressure) or electrocardiogram (ECG) parameters at Screening and check-in

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of APN1125 in healthy subjects via adverse events | 8 days
Assessment of safety and tolerability of APN1125 in healthy subjects via vital signs (e.g., blood pressure, pulse rate, respiratory rate, oral temperature) | 8 days
Assessment of safety and tolerability of APN1125 in healthy subjects via ECGs | 8 days
Assessment of safety and tolerability of APN1125 in healthy subjects via physical exams | 8 days
Assessment of safety and tolerability of APN1125 in healthy subjects via clinical laboratory tests (chemistry, hematology, coagulation and urinalysis) | 8 days

SECONDARY OUTCOMES:
Assessment of pharmacokinetics of APN1125 in plasma following single oral doses: maximum observed plasma concentration (Cmax) | 24 hours
Assessment of pharmacokinetics of APN1125 in plasma following single oral doses: time corresponding to occurrence of Cmax (tmax) | 24 hours
Assessment of pharmacokinetics of APN1125 in plasma following single oral doses: Area under the Curve from time zero to the last quantifiable concentration (AUClast) | 24 hours
Assessment of pharmacokinetics of APN1125 in plasma following single oral doses: Area under the Curve from time zero extrapolated to infinity (AUCinf) | 24 hours
Assessment of pharmacokinetics of APN1125 in plasma following single oral doses: terminal elimination rate constant (lz) | 24 hours
Assessment of pharmacokinetics of APN1125 in plasma following single oral doses: apparent elimination half-life (t1/2) | 24 hours
Assessment of pharmacokinetics of APN1125 in plasma following single oral doses: apparent plasma clearance (CL/F) | 24 hours
Assessment of pharmacokinetics of APN1125 in urine following single oral doses: apparent volume of distribution (Vz/F) | 24 hours
Assessment of pharmacokinetics of APN1125 in urine following single oral doses: urinary excretion (Ae) | 24 hours
Assessment of pharmacokinetics of APN1125 in urine following single oral doses: fraction of APN1125 dose excreted (Fe) | 24 hours
Assessment of pharmacokinetics of APN1125 in urine following single oral doses: urinary excretion expressed as percentage of dose administered (Ae%) | 24 hours
Assessment of pharmacokinetics of APN1125 in urine following single oral doses: renal clearance calculated as APN1125 (CLR) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: David Han, MD, Principal Investigator — California Clinical Trials Medical Group
Locations (1):
- PAREXEL Early Phase, Glendale, California, United States